CLINICAL TRIAL: NCT00630253
Title: A Study of Cyclophosphamide, Fludarabine, and Antithymocyte Globulin Followed by Matched Sibling Donor Hematopoietic Cell Transplantation in Patients With Fanconi Anemia
Brief Title: Cytoxan, Fludara, and Antithymocyte Globulin Conditioning Followed By Stem Cell Transplant in Treating Fanconi Anemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2000-09; 0001M34441 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-03-05; First posted 2008-03-06 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Fanconi Anemia
Keywords: Fanconi anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — Antilymphocyte Serum; Cyclophosphamide; fludarabine; fludarabine phosphate; Hematopoietic Stem Cell Transplantation; Methylprednisolone; Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Marrow Isolex (Experimental): bone marrow processed using Isolex 300i (for patients enrolled through April 2010)
  Interventions: Biological: Anti-Thymocyte Globulin; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Hematopoietic Stem Cell Transplantation; Drug: Methylprednisolone; Drug: Filgrastim; Drug: Cyclosporine; Drug: Mycophenolate Mofetil
- UCB (Experimental): No processing Notes: sibling donor UCB is used as the stem cell source and co-enroll for unlicensed UCB registry
  Interventions: Biological: Anti-Thymocyte Globulin; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Hematopoietic Stem Cell Transplantation; Drug: Methylprednisolone; Drug: Filgrastim; Drug: Cyclosporine; Drug: Mycophenolate Mofetil
- Marrow Clinimax (Experimental): bone marrow processed using CliniMACS (for patients enrolled beginning with the August 2010 protocol version)
  Interventions: Biological: Anti-Thymocyte Globulin; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Hematopoietic Stem Cell Transplantation; Drug: Methylprednisolone; Drug: Filgrastim; Drug: Cyclosporine; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin — 30 mg/kg/day will be administered after MP on days -6, -5, -4, -3 and -2.
  Other Names: ATG
Drug: Cyclophosphamide — 5 mg/kg is to be given as a 2 hour infusion, Days -6 through -3.
  Other Names: Cytoxan
Drug: Fludarabine — 35 mg/m^2 intravenously (IV) on days -6 through -2.
  Other Names: Fludara
Procedure: Hematopoietic Stem Cell Transplantation — Bone marrow or umbilical cord blood infusion on day 0.
  Other Names: HSCT
Drug: Methylprednisolone — Methylprednisolone (MP) 2 mg/kg/day intravenously every 24 hours will be given from day -6 until day -2 as a premedication for ATG.
  Other Names: MP
Drug: Filgrastim — 5 mcg/kg per day intravenously (IV) continue until Absolute neutrophil count > or = 2.5 x 10^9/L
  Other Names: G-CSF
Drug: Cyclosporine — Cyclosporine IV over 2 hours or orally every 8-12 hours beginning on day -3 and continuing until day 100, followed by a taper.
  Other Names: CSA
Drug: Mycophenolate Mofetil — Day -3 through day +30 or for 7 days after engraftment, whichever day is later, if no acute GVHD. Engraftment is defined as 1st day of 3 consecutive days of absolute neutrophil count [ANC] > 0.5 x 10^9/L. MMF will be given at a dose of 15 mg/kg/dose every 8 hours PO (to a maximum dose of 1 gram).
  Other Names: MMF

SUMMARY:
RATIONALE: Giving chemotherapy, such as cyclophosphamide and fludarabine, before a donor stem cell transplant helps to remove the patient's cells to allow for the transplant cells to take and grow. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells can make an immune response against the body's normal cells. Giving antithymocyte globulin and removing the T cells from the donor cells before transplant and giving cyclosporine before and after transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects of cyclophosphamide, fludarabine, and antithymocyte globulin followed by donor stem cell transplant and to see how well it works in treating patients with Fanconi anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the probability of engraftment in patients with Fanconi anemia treated with cyclophosphamide, fludarabine phosphate, and antithymocyte globulin followed by HLA-genotypically identical sibling donor hematopoietic stem cell transplantation that is T-cell depleted.

Secondary

* To evaluate the incidence of acute graft-versus-host disease (GVHD) and chronic GVHD in patients treated with this regimen.
* To evaluate the incidence of regimen-related toxicity in these patients.
* To evaluate the 1-year survival of patients treated with this regimen.
* To evaluate the incidence of late secondary malignancies (e.g., squamous cell carcinoma of the head and neck or cervix) in patients treated with this regimen.

OUTLINE:

* Preparative cytoreductive therapy: Patients receive cyclophosphamide IV over 2 hours on days -6 to -3 and fludarabine phosphate IV over 30 minutes and anti-thymocyte globulin IV over 4-6 hours on days -6 to -2.
* T-cell depleted donor hematopoietic stem cell transplantation: Patients undergo T-cell depleted donor bone marrow or umbilical cord blood stem cell transplantation on day 0. Patients also receive filgrastim (G-CSF) IV beginning on day 1 and continuing until blood counts recover.
* Graft-versus-host disease prophylaxis: Patients receive cyclosporine IV over 2 hours or orally every 8-12 hours beginning on day -3 and continuing until day 100, followed by a taper. Patients will receive Mycophenolate Mofetil (MMF) therapy beginning on day -3 through day +30 or for 7 days after engraftment, whichever day is later, if no acute GVHD. Engraftment is defined as 1st day of 3 consecutive days of absolute neutrophil count [ANC] > 0.5 x 10^9/L.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be <60 years of age with a diagnosis of Fanconi Anemia (FA).
* Patients must have an HLA-A, B, DRB1 identical sibling donor. Patients and donors will be typed for HLA-A and B using serological or molecular techniques and for DRB1 using high resolution molecular typing.
* Patients with FA must have moderately severe aplastic anemia (AA), early myelodysplastic syndrome (MDS) with no excess blasts with or without chromosomal abnormalities.

  * In patients <18 years of age, moderately severe aplastic anemia is defined as having at least one of the following:

    * platelet count <40 x 10^9/L
    * absolute neutrophil count (ANC) <10 x 10^8/L
    * Hgb <9 g/dL
  * In patients 18-60 years of age, moderately severe aplastic anemia is defined as having at least one of the following:

    * platelet count <20 x 10^9/L
    * absolute neutrophil count ANC <5 x 10^8/L
    * Hgb <8 g/dL
  * Early myelodysplastic syndrome, with multilineage dysplasia with < 5% blasts, with or without chromosomal anomalies.
* Adequate major organ function including:

  * Cardiac: ejection fraction >45%
  * Hepatic: no clinical evidence of hepatic failure (e.g. coagulopathy, ascites)
  * Karnofsky performance status >70% or Lansky >50%
* Women of child bearing age must be using adequate birth control and have a negative pregnancy test.

Exclusion Criteria:

* Active bacterial infection within one week of hematopoietic cell transplant (HCT)
* Active fungal infection at time of HCT.
* Late MDS with greater than 5% blasts in bone marrow.
* Acute myelogenous leukemia (AML) or history of AML
* Malignant solid tumor (e.g. squamous cell carcinoma of the head/neck/cervix) within 2 years of HCT.
* Pregnant or lactating female.

Max Age: 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2000-02-17 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L. MacMillan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Umbilical Cord Blood (UCB) Arm: No processing
Period: Overall Study
Arm/Group | Marrow Isolex | Umbilical Cord Blood (UCB) Arm | Marrow Clinimax
Started | 16 | 9 | 6
Completed | 16 | 9 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- UCB Arm: No processing
- Total: Total of all reporting groups
Arm/Group | Marrow Isolex | UCB Arm | Marrow Clinimax | Total
Number analyzed (Participants) | 16 | 9 | 6 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 9 | 4 | 26
  Between 18 and 65 years | 3 | 0 | 2 | 5
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 5 | 18
  Male | 7 | 5 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 8 | 6 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 12 | 7 | 3 | 22
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 9 | 6 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Graft Failure
Description: graft failure = absolute neutrophil count (ANC) <5 x 10^8/L and an acellular bone marrow aspirate/biopsy
Time Frame: From Day 1 to event, assessed up to100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | UCB Arm | Marrow Clinimax
Number analyzed (Participants) | 16 | 9 | 6
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Acute Graft-Versus-Host Disease (GVHD)
Description: Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | UCB Arm | Marrow Clinimax
Number analyzed (Participants) | 16 | 9 | 6
Participants | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Experiencing Overall Survival
Description: The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer. Also called survival rate.
  Overall survival will be defined as time from enrollment to date of death or censored at the date of last documented contact for patients still alive.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | UCB Arm | Marrow Clinimax
Number analyzed (Participants) | 16 | 9 | 6
Participants | 15 | 8 | 5

4. Secondary Outcome: Number of Participants With Chronic Graft-Versus-Host Disease (GVHD)
Description: Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | UCB Arm | Marrow Clinimax
Number analyzed (Participants) | 16 | 9 | 6
Participants | 2 | 0 | 0

5. Secondary Outcome: Number of Participants With Transplant Related Deaths
Description: In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | UCB Arm | Marrow Clinimax
Number analyzed (Participants) | 16 | 9 | 6
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Marrow Isolex | UCB Arm | Marrow Clinimax
All-Cause Mortality (participants affected / at risk) | 1/16 | 1/9 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/9 | 1/6
Other Adverse Events (participants affected / at risk) | 9/16 | 6/9 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marrow Isolex (N=16) | UCB Arm (N=9) | Marrow Clinimax (N=6)
Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — hemorrhage in the upper GI tract
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marrow Isolex (N=16) | UCB Arm (N=9) | Marrow Clinimax (N=6)
Brain Infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrect (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiopumonary shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Elevaed ALT (Investigations) | 2 (2) | 1 (1) | 0 (0)
Elevaed bilirubin (Investigations) | 1 (1) | 1 (1) | 0 (0)
GI bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Graft failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
Hypoxic ischemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 7 (27) | 5 (13) | 4 (10)
Intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Liver Ischemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ototoxicity (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pneumonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT00630253/Prot_SAP_000.pdf